CLINICAL TRIAL: NCT03285724
Title: Safety and Performance Study of the Harpoon Medical Device in Patients With Degenerative Mitral Regurgitation
Brief Title: Safety and Performance Study of the Harpoon Mitral Valve Repair System
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Edwards Lifesciences acquired Harpoon Medical in December 2017 and a decision has been made to close enrollment in the HMEFS-2000 protocol
Sponsor: Edwards Lifesciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HMEFS-2000
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Results first posted 2019-10-14 (Actual); Last update posted 2019-11-19 (Actual); Status verified 2019-11

CONDITIONS: Mitral Valve Regurgitation; Mitral Valve Prolapse; Mitral Valve Insufficiency
Keywords: Mitral Valve Repair; Transapical; artificial chordae; bi-leaflet prolapse; anterior prolapse; posterior prolapse
MeSH Terms: conditions — Mitral Valve Insufficiency; Mitral Valve Prolapse

STUDY DESIGN:
Intervention Model Description: Single Group Assignment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (1):
- Harpoon Medical Transapical device TSD-5 (Experimental): This is a prospective, single arm, nonrandomized, early feasibility study to evaluate the safety and performance of the Harpoon Medical Device.
  Interventions: Device: Harpoon Artificial ePTFE Chords

INTERVENTIONS:
Device: Harpoon Artificial ePTFE Chords — The Harpoon Medical Transapical device is intended to be used to reduce the degree of degenerative mitral regurgitation by delivering and anchoring one or more ePTFE cords to the affected mitral valve leaflet(s) via a small left thoracotomy on the beating heart in patients with anterior, bi-leaflet or posterior prolapse.

SUMMARY:
The primary objective of this study is to evaluate the safety and performance of the Harpoon Medical Device. It is anticipated, that the Harpoon Medical Device will provide advantages over current surgical interventions including: 1) a small minimally invasive incision, 2) no sternotomy, 3) no cardiopulmonary bypass, 4) no aortic manipulation, 5) a direct path to the valve plane, 6) performed on a beating heart, 7) real-time TEE-guided ePTFE cordal length adjustment and 8) less complicated procedure that is teachable and adoptable.

DETAILED DESCRIPTION:
The device is designed to reduce the degree of mitral regurgitation by delivering and anchoring artificial chordae tendineae to the affected mitral valve leaflet(s) in a beating heart.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient referred for mitral valve surgery
* Presence of severe MR as read on an echocardiographic study performed within 60 days prior to procedure.
* Estimated post-ePTFE cordal implantation coaptation surface is adequate in the judgment of the operating surgeon and the patient eligibility committee
* Degenerative mitral valve disease associated with anterior, bileaflet, or posterior leaflet prolapse
* Patient is able to sign informed consent and able to return for follow-up and is capable of participating in all testing associated with this clinical investigation
* Women of child-bearing potential have a negative pregnancy test

Exclusion Criteria:

* Age < 18 years
* Infective endocarditis
* History of Mediastinal Radiation
* Inflammatory (rheumatic) valve disease
* Requirement for concomitant cardiac surgery (e.g., coronary artery bypass grafting (CABG), aortic valve surgery, etc.)
* Symptomatic coronary artery disease
* Cardiogenic shock at the time of enrollment
* ST segment elevation myocardial infarction requiring intervention within 30 days prior to enrollment
* Evidence of cirrhosis or hepatic synthetic failure
* Pregnancy at the time of enrollment (women of child bearing age should have negative pregnancy within 14 days of surgery)
* Severe pulmonary hypertension (PA systolic pressure > 70 mmHg)
* Previous cardiac surgery, or surgery on the left pleural space
* Left ventricular, atrial or appendage thrombus
* Severely calcified mitral leaflets
* Recent stroke (< 6 months) with permanent impairment
* EuroScore (for mitral valve repair) > 8%
* Patients with contraindications to Transesophageal echocardiography
* Severe left or right ventricular dysfunction
* NYHA Class IV
* Renal insufficiency CKD stage 3b or worse (GFR < 45 ml/min/1.73 m2)
* Patient is participating in another clinical study for which follow-up is currently ongoing. (Co-enrollment in an investigational device or interventional study)
* Patient with non-cardiac co-morbidities and life expectancy < 1 year
* Patient has a condition or conditions that, in the opinion of the Investigator, preclude participation, including willingness to comply with all follow-up procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2017-05-16 (Actual); Primary Completion 2017-06-16 (Actual); Study Completion 2018-04-20 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Bartus, MD PhD, Principal Investigator — Jagiellonian University
Locations (2):
- Poland (2):
  - Jagiellonian University, Krakow
  - Instytut of Kardiologii & Transplantology, Warsaw

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Harpoon Medical Device: Safety and Performance study of the Harpoon Medical Device in patients with degenerative mitral regurgitation.
Period: Overall Study
Arm/Group | Harpoon Medical Device
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Harpoon Medical Device
Number analyzed (Participants) | 1
Age, Customized [Number; unit: years]
  Age | 70
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Subjects With Procedural Success During the First 30 Days
Description: To demonstrate that the Harpoon Medical Device performs as designed and can successfully implant one or more ePTFE artificial cords on either the anterior, posterior, or both leaflets of the mitral valve via a small left thoracotomy on the beating heart and reduce mitral regurgitation from "severe" to less than or equal to "moderate" at the conclusion of the procedure and at 30 days post-procedure.
Time Frame: Procedure, discharge, and 30 days
Population: Subject was not implanted with study Device
Measure: Count of Participants; unit: Participants
Arm/Group | Harpoon Medical Device
Number analyzed (Participants) | 1
Participants
  Procedure | 0
  Discharge | 0
  30 days follow-up | 0

2. Primary Outcome: Number of Subjects With Freedom From Serious Adverse Events (SAE) During the First 30 Days
Description: Procedure freedom from Serious Adverse Events (SAEs) during the procedure, at discharge, and at 30 days follow-up shall be tracked and recorded.
Time Frame: Procedure, Discharge and 30 Days
Measure: Count of Participants; unit: Participants
Arm/Group | Harpoon Medical Device
Number analyzed (Participants) | 1
Participants
  Procedure | 0
  Discharge | 0
  30 Days | 0

3. Secondary Outcome: Subject's Severity of Mitral Regurgitation Over Time
Description: Severity of mitral regurgitation at 6 months, 12 months and 24 months follow-up shall be tracked and recorded
Time Frame: 6 Months, 12 Months, and 24 Months
Population: Participant did not receive the Harpoon Medical Device.
Arm/Group | Harpoon Medical Device
Number analyzed (Participants) | 0

4. Secondary Outcome: Subject's Freedom From Serious Adverse Events Over Time
Description: Freedom from Serious Adverse Events (SAEs) at 6 months, 12 months and 24 months follow-up shall be tracked and recorded
Time Frame: 6 Months, 12 Months, and 24 Months
Population: Participant did not receive the Harpoon Medical Device.
Arm/Group | Harpoon Medical Device
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: Events occurring from baseline through end of procedure.
Description: Participant did not receive the Harpoon Medical Device.
Arm/Group | Harpoon Medical Device
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 0/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Harpoon Medical Device (N=1)
Implantation cord failure, mitral ring damage (Cardiac disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
PI must submit publication 60 days prior to its submission for presentation/publication to Sponsor. The Sponsor may, at its sole discretion, (a) approve the publication, (b) reject the publication, or (c) suggest changes to the publication to ensure protection of confidential commercial information in compliance with regulatory requirements. Until the content of any publication is approved by the Sponsor and the PI, the PI shall not disclose such publication.

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2016-10-12): https://cdn.clinicaltrials.gov/large-docs/24/NCT03285724/Prot_SAP_000.pdf